CLINICAL TRIAL: NCT04153461
Title: Mini- Percutaneous Nephrolithotomy Versus Standard Percutaneous Nephrolithotomy in the Treatment of Renal Stones. A Randomized Controlled Trial
Brief Title: Mini- Percutaneous Nephrolithotomy Versus Standard Percutaneous Nephrolithotomy in the Treatment of Renal Stones.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa Elgamal, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MiniPNL
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Urolithiasis; Stone;Renal; Nephrolithiasis; PNL; PCNL; NEPHROLITHOTOMY; MINIPERC
Keywords: urolithiasis; stone, renal; nephrolithiasis; PNL; PCNL; NEPHROLITHOTOMY; MINIPERC; MINI-PERC; BLOOD LOSS; NEPHROSTOMY SIZE
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINI-PERCUTANEOUS NEPHROLITHOTOMY (Active Comparator): MINIPERCUTANEOUS NEPHROLITHOTOMY USING NEPHROSCOPY 15 FR, LASER DUSTING OF THE STONE, NEPHROSTOMY TUBE 12 FIXATION
  Interventions: Procedure: MINI-PERCUTANEOUS NEPHROLITHOTOMY
- STANDARD PERCUTANEOUS NEPHROLITHOTOMY (Active Comparator): PERCUTANEOUS NEPHROLITHOTOMY USING NEPHROSCOPY 24 FR, ULTRASOUND OR LITHOCLAST DISINTEGRATION OF THE STONE AND FORCEPS EXTRACTION OF THE FRAGMENTS, NEPHROSTOMY TUBE 22 FIXATION
  Interventions: Procedure: STANDARD PERCUTANEOUS NEPHROLITHOTOMY

INTERVENTIONS:
Procedure: MINI-PERCUTANEOUS NEPHROLITHOTOMY — MINIPERCUTANEOUS NEPHROLITHOTOMY USING NEPHROSCOPY 15 FR, LASER DUSTING OF THE STONE, NEPHROSTOMY TUBE 12 FIXATION
  Other Names: MINIPERC; MINI-PERC
  Arms: MINI-PERCUTANEOUS NEPHROLITHOTOMY
Procedure: STANDARD PERCUTANEOUS NEPHROLITHOTOMY — PERCUTANEOUS NEPHROLITHOTOMY USING NEPHROSCOPY 24 FR, ULTRASOUND OR LITHOCLAST DISINTEGRATION OF THE STONE AND FORCEPS EXTRACTION OF THE FRAGMENTS, NEPHROSTOMY TUBE 22 FIXATION
  Other Names: PNL; PCNL; STANDARD PNL
  Arms: STANDARD PERCUTANEOUS NEPHROLITHOTOMY

SUMMARY:
The EUA Urolithiasis Guidelines Panel meta-analysis suggest that mPNL is at least as efficacious and safe as sPNL for the removal of renal calculi. However, the quality of the evidence was poor, drawn mainly from small studies, the majority of which were single-arm case series, and only one of which was RCT. The risks of bias and confounding were high, highlighting the need for more reliable data from RCTs. So, the Panel recommended for more clinical research .

The aim of this study is to compare between PNL and mPNL through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 18 years or older.
2. ASA I or II
3. Renal stones ≥ 2 cm
4. Lower calyceal stone ≥ 1 cm
5. Failure of other modalities of treatment as ESWL and RIRS.

Exclusion Criteria:

1. S.creatinine > 2mg/dl.
2. Patients with active UTI.
3. Patients on anticoagulant.
4. Age <18 years.
5. Ureteral obstruction preventing the insertion of a ureteral stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of stone free rate (SFR) | 2 years
  defined as less than 4mm by non contrast computed tomography

SECONDARY OUTCOMES:
assessment of haemoglobin loss | 2 years
  measured by haemoglobin change pre and postoperative (measured by grams/ deciliter)
assessment of pain | 2 years
  measured by visual analogue scale
assessment of renal function | 2 years
  measured by serum creatinine measured by Milligram/ deciliter
assessment of patient satisfaction | 2 years
  measured by freiburg index of patient satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: No